CLINICAL TRIAL: NCT04195932
Title: Exercise as a Modulator of Immune Risk Factors for Ischemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, John Kelly Smith, Emeritus Professor of Medicine, East Tennessee State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ETSU2
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Heart Diseases
Keywords: exercise; hyperlipidemia; TNF-alpha; atherogenesis; LDL-cholesterol; oxidized LDL-C
MeSH Terms: conditions — Heart Diseases; Motor Activity; Hyperlipidemias; Atherosclerosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Before and after study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): 6 moths of supervised moderate intensity aerobic and resistive exercise training
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training

SUMMARY:
A before and after study involving 43 adult subjects at risk of having ischemic heart disease. Subjects underwent 6 months of supervised moderate intensity aerobic and resistive exercise training. Blood samples were obtained at entry and at 6 months for measurement of complement (C3), CRP, blood lipid levels, lymphocyte phenotypes, and for the isolation, culture, and measurement of the spontaneous and phytohemagglutinin-induced secretion of proatherogenic and antiatherogenic cytokines by their peripheral blood mononuclear cells (PBMC).

DETAILED DESCRIPTION:
A before and after study involving 43 adult subjects at risk of having ischemic heart disease. Subjects underwent 6 months of supervised moderate intensity aerobic and resistive exercise training. Blood samples were obtained at entry and at 6 months for measurement of complement (C3), CRP, blood lipid levels, lymphocyte phenotypes, and for the isolation, culture, and measurement of the spontaneous and phytohemagglutinin-induced secretion of proatherogenic and antiatherogenic cytokines by their peripheral blood mononuclear cells (PBMC

ELIGIBILITY:
Inclusion criteria:

* normal EKG
* normal stress test

Exclusion Criteria:

* abnormal EKG
* abnormal stress test
* presence of a chronic inflammatory disease
* presence of malignancy
* immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 1996-12 (Actual); Primary Completion 1998-05 (Actual); Study Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Effect of exercise on atherogenic cytokine production by mitogen-stimulated peripheral blood mononuclear cells | 1 year
  Pre- and post-exercise peripheral blood mononuclear cell (PBMC) preparations are isolated from venous blood, washed three times at 10 degrees C with sterile phosphate buffered saline (pH 7.4, 0.1 M) and suspended at a concentration of 2 million cells/uL in RPMI-1640. Preparations are incubated under 5% CO2 at 37 degrees C for 48 hours with phytohemagglutinin (5 ug/ml). Culture supernatants are rendered cell-free and supernatants assayed for Interleukin (IL)-1α, tumor necrosis factor (TNF)-α, and interferon (IFN)-γ using solid phase enzyme linked immunoassay kits.
Effect of exercise on plasma lipids and oxidizable low density lipoprotein cholesterol levels | 1 year
  Pre- and post-exercise fasting plasma levels of total cholesterol (TC), very low density lipoprotein cholesterol (VLDL), low density lipoprotein cholesterol (LDL-C), and high density lipoprotein cholesterol (HDL-C) levels are measured using g-Max Quick-Seal tubes and potassium bromide (KBr) (d=1.006 g/mL). Tubes are centrifuged for 120 minutes at 68,000 rpm at 14 degrees C. The top layer (VLDL) is harvested, the bottom 3.7 mL adjusted to a density of 1.063 g/mL with KBr, and the tubes centrifuged for 150 minutes at 68,000 rpm at 14 degrees C to float the LDL-C. The bottom layer contains the HDL-C. TC, VLDL-C, LDL-C, and HDL concentrations are measured colorimetrically. LDL oxidizability is measured by oxidizing LDL-C (0.05 g/L) with 50 ug/mL Cu++ at 30 degrees C and measuring diene levels spectrometrically at 234 nm.

SECONDARY OUTCOMES:
Effect of exercise on blood lymphocyte phenotypes | 1 year
  Pre- and post-exercise blood samples are immunophenotyped using lysed whole blood, a FACScan flow cytometer, and fluorescein- and phycoerythrin-labeled murine monoclonal IgG antibodies to measure levels of T lymphocytes (CD3+), T helper lymphocytes (CD4+), T cytotoxic lymphocytes (CD8+), and T lymphocytes displaying MHC class II antigen (DR+), vascular adhesion molecule-4 (VLA-4) (CD49d+), lymphocyte function-associated antigen-1 (LFA-1) (CD11a+), Fas antigen (CD95+), and gamma-delta T cell receptors (TCR gamma-delta+). Also measured are B lymphocytes (CD3-CD19+), B1 lymphocytes (CD3-CD19+CD5+) and natural killer cells (NK cells) (CD3-CD16+CD56+).

CONTACTS AND LOCATIONS:
Overall Officials: John K Smith, MD, Principal Investigator — East Tennessee State University
Locations (1):
- James H. Quillen College of Medicine, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No